CLINICAL TRIAL: NCT04975958
Title: An Open-Label, Multicenter, Phase 1a Study of AN2025 and AN0025 in Double Combination With Atezolizumab and in Triple Combination With Atezolizumab in Patients With Advanced Solid Tumors
Brief Title: Double/Triple Combinations of AN2025, AN0025 and Atezolizumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adlai Nortye Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN2025S0101
Record Dates: First submitted 2021-07-02; First posted 2021-07-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Solid Tumor
MeSH Terms: interventions — NVP-BKM120; E7046; atezolizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DLT Observation Period I - AN2025 and Atezolizumab (Experimental): During the DLT Observation I, patients will be treated with AN2025 and Atezolizumab until the patient experiences disease progression, unacceptable toxicity or withdraws consent. The starting dose of AN2025 is 50 mg. If tolerated, then a subsequent cohort will escalate to 100 mg. A dose de-escalation cohort to 80 mg may occur if the 100 mg is not well tolerated. The dose of Atezolizumab will remain constant at 1200 mg every 3 weeks (Q3W) for each dose level of AN2025 and in each cohort. Atezolizumab is administered intravenously over 60 minutes. If the first infusion is tolerated, all subsequent infusions may be delivered over 30 minutes.
  Interventions: Drug: AN2025; Drug: Atezolizumab 1200 mg in 20 ML Injection
- DLT Observation Period II - AN0025 and Atezolizumab (Experimental): During the DLT Observation II, patients will be treated with AN0025 and Atezolizumab until the patient experiences disease progression, unacceptable toxicity or withdraws consent. The starting dose of AN0025 is 250 mg. If tolerated, then a subsequent cohort will escalate to 500 mg. If 250 mg AN0025 is not tolerated, de-escalate to 125 mg. The dose of Atezolizumab will remain constant at 1200 mg Q3W for each dose level of AN0025 and in each cohort. Atezolizumab is administered intravenously over 60 minutes. If the first infusion is tolerated, all subsequent infusions may be delivered over 30 minutes.
  Interventions: Drug: AN0025; Drug: Atezolizumab 1200 mg in 20 ML Injection
- DLT Observation Period III - AN2025, AN0025 and Atezolizumab (Experimental): The DLT Observation III will be started after safety data review by the investigators and the sponsor of the double combination treatments in Observations I and II. Patients enrolled in Observation III will start with the recommended dose of AN0025 from Observation II, 1200 mg Atezolizumab, and AN2025 will start from 50 mg QD. Patients will be treated with all three study drugs until the patient experiences disease progression, unacceptable toxicity or withdraws consent. The dose of Atezolizumab will be the same (i.e., 1200 mg Q3W) regardless of dose levels of AN2025 and cohorts. Atezolizumab is administered intravenously over 60 minutes every three weeks. If the first infusion is tolerated, all subsequent infusions may be delivered over 30 minutes. The dose of AN0025 as determined in Observation II will remain constant for each dose level of AN2025 and each cohort, unless the investigators and the sponsor determine that the toxicity comes from the AN0025 + Atezolizumab combination.
  Interventions: Drug: AN2025; Drug: AN0025; Drug: Atezolizumab 1200 mg in 20 ML Injection

INTERVENTIONS:
Drug: AN2025 — oral administration
  Other Names: BKM120
  Arms: DLT Observation Period I - AN2025 and Atezolizumab; DLT Observation Period III - AN2025, AN0025 and Atezolizumab
Drug: AN0025 — oral administration
  Other Names: E7046
  Arms: DLT Observation Period II - AN0025 and Atezolizumab; DLT Observation Period III - AN2025, AN0025 and Atezolizumab
Drug: Atezolizumab 1200 mg in 20 ML Injection — infusion
  Other Names: Tecentriq

SUMMARY:
This is an open-label, multicenter, Phase 1a study to evaluate the safety, tolerability, PK and preliminary efficacy of AN2025 and AN0025 in double or triple combination treatments with Atezolizumab in patients with locally advanced/metastatic tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1a study to evaluate the safety, tolerability, PK and preliminary efficacy of AN2025 and AN0025 in double or triple combination treatments with Atezolizumab in patients with locally advanced/metastatic tumors. This study consists of three DLT Observation Periods I, II and III. Observations I and II are double combination treatments, which will be conducted in parallel, whereas Observation III (the triple combination treatment) will be initiated only after a thorough review of the safety data from Observations I and II. In all three Observation Periods, a "6 + 3 design" will be utilized for dose finding with dose escalation and de-escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of informed consent and have provided signed informed consent for the trial.
2. Willing and able to comply with all aspects of the protocol.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Life expectancy ≥3 months.
5. Diagnosed with histologically confirmed locally advanced and nonresectable, or metastatic disease.
6. Have received at least one line of prior systemic therapy or no alternative therapy to prolong survival exists.
7. Have received no more than 4 prior lines of systemic therapy for advanced disease. Prior therapy in an adjuvant or neoadjuvant setting is not considered as a prior line of systemic therapy.
8. Have measurable disease per RECIST 1.1 as assessed by the local site investigator and/or radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
9. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. If previously treated with anti-PD-1/PD-L1 therapy, tumor tissue sample obtained following the most recent anti-PD-1/PD-L1 therapy is required. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
10. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple gated acquisition (MUGA) scan.
11. Patient has organ function as shown by the following:

    1. Absolute neutrophil count (ANC) ≥1.5 x 109/L.
    2. Hemoglobin ≥9 g/dL (which may be reached by transfusion 2 weeks prior to the start of the study treatment).
    3. Platelets ≥100 x 109/L (which may be reached by transfusion).
    4. International normalized ratio (INR) ≤1.5.
    5. Calcium (corrected for serum albumin) within normal limits (WNL) or ≤ grade 1 severity according to NCI-CTCAE version 5.0 if judged clinically not significant by the Investigator. Patients concomitantly taking bisphosphonates or denosumab for calcium correction are eligible. (only applicable to Observations I and III)
    6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x upper limit of normal (ULN) or <5.0 x ULN if liver metastases are present.
    7. Total serum bilirubin ≤ ULN or ≤1.5 x ULN if liver metastases are present; or total bilirubin ≤3.0 x ULN with direct bilirubin below or within normal range in patients with well documented Gilbert's Syndrome. Gilbert's syndrome is defined as presence of episodes of unconjugated hyperbilirubinemia with normal results from cells blood count (including normal reticulocyte count and blood smear), normal liver function test results, and absence of other contributing disease processes at the time of diagnosis.
    8. Serum creatinine ≤1.5 x ULN or calculated or directly measured creatinine clearance (CrCL) >30 mL/min.
    9. HbA1c ≤8%. (Only applicable to Observations I and III)
12. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks prior to Screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment, is she considered not of child-bearing potential.
    2. Woman of childbearing potential who agrees to follow contraceptive guidance during the treatment period and for at least 5 months after the last dose of Atezolizumab.

    Highly effective contraception is defined as either:
    * Total abstinence: When this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
    * Female sterilization: When the female study patient has had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female study patients, the vasectomized male partner should be the sole partner for that patient.
    * Using a combination of any two of the following:

      * Placement of an intrauterine device (IUD) or intrauterine system (IUS), and
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
      * Hormonal contraception methods (e.g., oral, injected, implanted).
13. A male participant must agree to use contraception during the treatment period and for at least 5 months after the last dose of Atezolizumab.

Exclusion Criteria:

1. Have been discontinued treatment due to a Grade 3 or higher immune-related AE (irAE) from prior anti-PD-1or anti-PD-L1, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
2. Have received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives, whichever is shorter.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or returned to baseline. Participants with ≤ Grade 2 neuropathy or alopecia may be eligible.
3. Have received prior palliative radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
4. Severe, uncontrolled tumor-related pain.
5. Have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Non live COVID vaccinations or boosters should not occur during Cycle 1 or within 30 days prior to the first dose of study drug.
6. Are currently participating in a study of an investigational agent or have used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been at least 4 weeks after the last dose of the previous investigational agent (see Number 2 above).
7. Have had an allogenic tissue/solid organ transplant.
8. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
9. With a history of another primary malignancy within the past 2 years, with the exception of basal or squamous cell skin cancer, or carcinoma in situ of the cervix or breast that has undergone potentially curative therapy.
10. Have known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
11. Have known severe hypersensitivity to study treatment components.
12. Have an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed. Have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis.
13. Have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis.
14. Have an active infection requiring systemic therapy within 2 weeks prior to Day 1 of Cycle 1.
15. Participants with known human immunodeficiency virus (HIV) and/or history of Hepatitis B or C infections, or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) DNA or Hepatitis C Antibody or RNA. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
16. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment (including oral anticoagulation).
17. Major surgery within 4 weeks before the first dose of study drug. Note: If participant received major surgery, they must have recovered adequately from surgery and the toxicity and/or complications requiring the intervention prior to starting study treatment.
18. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the oral bioavailability of the investigational drugs.
19. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
20. Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study, e.g. history of or active major depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia, or history of suicidal attempt or ideation, homicidal ideation (e.g., risk of doing harm to self or others), or patients with active severe personality disorders (defined according to Diagnostic and Statistical Manual of Mental Disorders [DSM V]) are not eligible. Note: For patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous six weeks prior to start of study drug.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 5 months after the last dose of Atezolizumab.
22. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures >/=1 time per month.
23. Leptomeningeal disease.
24. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated but without evidence that disease has been clinically stable for >/=2 weeks prior to Day 1 of Cycle 1.
25. Oral or IV antibiotics within 2 weeks prior to Day 1 of Cycle 1 for an active infection (prophylactic antibiotic dosing that is deemed to be essential by the investigator is allowed).
26. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
27. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation.
28. Active tuberculosis.
29. Patient has received previous treatment with any protein kinase B (PKB/AKT), mammalian target of rapamycin (mTOR) inhibitors, or phosphatidylinositol 3 kinase (PI3K) pathway inhibitors (only applicable to Observations I and III).
30. Patient has grade ≥2 neuropathy, colitis, pneumonitis, elevated HbA1C, and uncontrolled endocrinopathies (e.g., hypothyroidism) from previous treatment (only applicable to Observations I and III).
31. Have clinically manifest diabetes mellitus (DM) (treated and/or with clinical signs) that is not well controlled (only applicable to Observations I and III).
32. Patient is currently receiving warfarin or other coumarin-derived anti-coagulant, or anti-Xa agents, for treatment, prophylaxis, or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), fondaparinux or novel oral anticoagulants (NOACs) is allowed.
33. Have diarrhea ≥2 CTCAE Grade 2 (only applicable to Observations I and III).
34. Patient is currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A4, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug (only applicable to Observations I and III). UGT inducers or inhibitors such as atazanavir, probenecid, valproic acid, mefenamic acid, quinidine (only applicable to Observation II).
35. Patient has a history of non-compliance to any medical regimen or inability to grant consent.
36. Patient that is currently receiving NSAIDs.
37. Patient that is currently receiving angiotensin converting enzyme (ACE) inhibitors and angiotensin II receptor blockers (ARBs): Patients on these hypertensives at study entry should be switched to other hypertensives prior to study drug dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure - Dose Limiting Toxicities (DLTs) | 3 weeks
  Number of participants with Dose Limiting Toxicities (DLTs)
Primary Outcome Measure - Number of participants with adverse events and serious adverse events | 2 years
  The safety profile will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0

SECONDARY OUTCOMES:
Overall Response Rate (ORR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 2 years
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR), by Investigator review and in accordance with RECIST 1.1.
Progression-Free Survival (PFS) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 2 years
  PFS is defined as the time from the date of the first dose of study drug to the date of the first documentation of disease progression or death, whichever occurs first.
Duration of Response (DOR) | 2 years
  DOR is defined as the time from the earliest objective response to disease progression or death.
Overall Survival (OS) | 2 years
  OS is defined as the time from the date of the first dose of study drug to the date of death.
Efficacy by Phosphatidylinositol-4,5-bisphosphate 3 Kinase Catalytic Subunit Alpha (PIK3CA) mutation in DLT Observations I and III | 2 years
  Efficacy by PIK3CA mutation in Observation I and III

CONTACTS AND LOCATIONS:
Overall Officials: Robert Atkinson, PhD, MSCR, Study Director — Adlai Nortye US Inc
Locations (5):
- United States (5):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Cancer Specialists - Lake Mary Cancer Center, Lake Mary, Florida
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Grossman School of Medicine, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No